CLINICAL TRIAL: NCT00953589
Title: 480 STUDY: Phase 2b Open-label, Randomized Study in Treatment Naïve Subjects With HCV G1 to Compare the Efficacy, Safety, and Tolerability of the 480 µg Dose of Locteron™ Plus Ribavirin Given Bi-Weekly to PEG-Intron™ Plus Ribavirin Given Weekly
Brief Title: 480 STUDY: Phase 2b Study of Locteron Plus Ribavirin to Treat Hepatitis C Virus (HCV)
Acronym: 480S
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biolex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLX883-204
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C, Chronic
Keywords: treatment naive
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Locteron ® PANEL A (Experimental): PANEL A: Locteron™ 480 µg dosed every 2 weeks in two subcutaneous injections (160 µg and 320 µg)
  Interventions: Drug: ribavirin
- Locteron ® PANEL B (Experimental): PANEL B: Locteron™ 480 µg dosed every two weeks in single subcutaneous injections
  Interventions: Drug: ribavirin
- PEG-Intron® PANEL A (Active Comparator): PEG-Intron® 1.5 µg/kg body weight weekly subcutaneous injection
  Interventions: Drug: ribavirin
- PEG-Intron® PANEL B (Active Comparator): PEG-Intron® 1.5 µg/kg body weight weekly subcutaneous injection
  Interventions: Drug: ribavirin

INTERVENTIONS:
Drug: ribavirin — Ribavirin - oral administration Subjects with body weight < 65 kg: 800 mg/day Subjects with body weight 65-85 kg: 1000 mg/day Subjects with body weight 86-105 kg: 1200 mg/day Subjects with body weight > 105 kg: 1400 mg/day
  Other Names: Ribasphere

SUMMARY:
The purpose of this 12-week study was to assess in subjects with chronic hepatitis C (treatment-naïve, genotype 1) receiving weight-based doses of ribavirin the early virologic response to the 480 ug dose level of Locteron™, dosed every 2 weeks, in comparison with 1.5 ug/kg PEG-Intron™ dosed weekly.

DETAILED DESCRIPTION:
The aim of the 480 STUDY was to compare efficacy and safety of 480ug Locteron dosed every other week to 1.5 ug/kg PegIntron dosed weekly in treatment-naïve genotype-1 chronic HCV subjects treated with weight-based ribavirin. This 12-week study was comprised of two panels (Panel A and Panel B). The designs of both panels were identical. HCV RNA was measured weekly for three weeks and then every other week. Adverse events including flu-like events and depression were collected during weekly clinic visits for 12 weeks. Flu-like events were also collected daily for 12 weeks by subject self-report using the internet (ePRO). Beck Depression Inventory (BDI) and Short Form-36 scores were measured at baseline and monthly through Week 12.

In Panel A of 480 STUDY, 42 treatment-naïve subjects with chronic genotype-1 HCV in Bulgaria and Romania were randomized and dosed with either Locteron q2weeks or weekly PegIntron, both in combination with weight-based ribavirin (13). In Panel A, 19 subjects received 480ug Locteron and 23 subjects received PegIntron.

In Panel B of 480 STUDY, 32 treatment-naïve subjects with genotype-1 HCV in Israel were randomized and dosed with either Locteron q2weeks or weekly PegIntron, both in combination with weight-based ribavirin (13). In Panel B, 16 subjects received 480ug Locteron and 16 subjects received PegIntron.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 through 69 years of age, inclusive
* Chronic hepatitis C genotype 1
* HCV ribonucleic acid (RNA) level > 10,000 IU/mL (by RT-PCR) at screening
* Creatine clearance ≥ 50 mL/min
* Neutrophil count > 1500 cells/mm3
* Platelet count > 90,000/mm3
* Hemoglobin > 12 g/dL for females and > 13 g/dL for males
* Female subjects of child-bearing potential agreeing to use dual methods for contraception
* Male subjects with female sexual partners agreeing to use effective birth control methods
* Negative serum pregnancy test for women of child-bearing potential
* Compensated liver disease defined as INR < 1.5, conjugated bilirubin < 1.5 x ULN, serum albumin > 3.0 g/dL
* Histologic evidence of Chronic Hepatitis C (CHC) (inflammation, fibrosis and/or cirrhosis on a standardized histologic grading system) as shown by biopsy within 2 years of screening or agrees to have a liver biopsy performed prior to randomization.

Exclusion Criteria:

* Prior antiviral treatment for hepatitis C
* Co-infection with HIV or hepatitis B virus
* Subjects with a body mass index (BMI) above 32 kg/m2
* Current or prior history of clinical hepatic decompensation
* Evidence of HCC
* Uncontrolled diabetes mellitus as evidenced by HbA1C ≥ 8.5% at screening
* Known hypersensitivity to interferon alfa or ribavirin
* Chronic liver disease other than HCV
* Clinically significant hemoglobinopathy
* History of moderate, severe or uncontrolled psychiatric disease including depression and prior suicide attempts
* History of immune-mediated disease
* Significant renal or neurological disease
* Severe degree (> GOLD stage III) of chronic pulmonary disease (COPD) or active, severe asthma
* Subjects with severe cardiac disease
* History of significant central nervous system (including CNS trauma) or seizure disorders
* Cancer within the last 5 years, or previous cancer with a high risk of recurrence
* History of solid organ or bone marrow transplantation
* Clinical or laboratory evidence of uncontrolled thyroid disease, e.g., by thyroid stimulating hormone (TSH) level > 1.2 x upper limit of normal
* Clinically significant retinopathy; this needs to have been excluded by an eye exam performed by an ophthalmologist within the last 6 months prior to screening for subjects with hypertension or diabetes mellitus
* Drug abuse or alcohol consumption within the last 6 months which, in the opinion of the investigator, may affect study participation or outcome. Subjects in a supervised methadone treatment program on a stable regimen for > 6 months may be considered
* Taken any experimental agent within 12 weeks prior to screening
* More than 30 days of systemic immunosuppressive medication to include steroids in doses equivalent to or greater than 10 mg prednisone per day within 30 days prior to screening (inhaled corticosteroids are allowed)
* Nursing mother or male partner of pregnant female.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: EVR: the proportion of subjects in each arm that have at least a 2 log drop in HCV RNA from Baseline | Week 12

SECONDARY OUTCOMES:
the proportion of subjects in each arm demonstrating HCV RNA undetectable (< 10 IU/mL) after 12 weeks of randomized treatment | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Walker A. Long, MD, Study Director — Biolex Therapeutics
Locations (15):
- Bulgaria (6):
  - Tokuda Hospital, Sofia
  - UMHAT "Alexandrovska", Sofia
  - UMHAT "St Ivan Rilski", Sofia
  - UMHAT "Queen Giovanna - ISUL" EAD, Sofia
  - Medical Institute Ministry of Interior, Sofia
  - UMHAT "St Maria", Varna
- Israel (5):
  - Carmel Medical Center, Haifa
  - Holy Family Hospital Nazareth, Nazareth
  - Rabin Medical Center, Petah Tikva
  - Rebekah Ziv Medical Center Safed, Safed
  - Sourasky Medical Center, Tel Aviv
- Romania (4):
  - Institute of Infectious Diseases, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - "Victor Babes" Clinical Hospital Craiova, Craiova
  - Gastroenterology and Hepatology Institute, Iași

REFERENCES:
- [Background] Krastev Z, Kotzev I, Tchernev K, Rigney A, Nikolovska D, Vladimirov B, Caruntu FA, Diaconescu IG, Voiculescu XX, Long, WA. Randomized, open-label, 12-week comparison of controlled-release interferon alpha2b + ribavirin vs. pegylated interferon alpha 2b +ribavirin in treatment-naïve genotype1 hepatitis C: 4 week results from 480STUDY (Panel A). J Hepatology 52:S27 (abstract 58), 2010. (Presented to 45th Annual Meeting of the European Association for the Study of the Liver, April 16, 2010, Vienna, Austria.)